CLINICAL TRIAL: NCT00106197
Title: Treatment Prediction in Adolescent and Adult Depression
Brief Title: Hormone and Sleep Response to Antidepressant Treatment in Adolescents and Adults With Depression
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Uma Rao (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Uma Rao, Principal investigator, Meharry Medical College
Organization: Meharry Medical College (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01MH068391 (NIH); DDTR B4-ARD; R01MH068391 (NIH)
Record Dates: First submitted 2005-03-21; First posted 2005-03-22 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Depression
Keywords: Sleep, REM; Antidepressant; Adolescent; Cortisol
MeSH Terms: conditions — Depression | interventions — Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Participants will receive bupropion in the sleep study
  Interventions: Drug: Bupropion

INTERVENTIONS:
Drug: Bupropion — Participants will start with 150 mg daily. If no adverse symptoms, dosage will be increased to twice daily. Treatment will last for 8 weeks.

SUMMARY:
This study will determine whether there are age-related differences in the body systems controlling sleep and stress hormone patterns. This study will also determine whether the differences in sleep and hormone patterns between depressed adolescents and adults are associated with differences in their response to antidepressant treatment.

DETAILED DESCRIPTION:
Adolescent depression is a serious public health concern that may lead to functional disability and death. The problems associated with the condition may continue into adulthood; therefore, early identification and effective treatment of adolescent depression is critical. Studies indicate that depressed adolescents experience greater variations in sleep and hormone patterns than depressed adults. These variations may influence responses to antidepressant treatment. This study will examine the mechanisms underlying developmental differences in sleep and hormone patterns to develop a strategy for identifying adolescents and adults who could benefit from antidepressant treatment.

This study will last approximately 10 weeks. At study start, participants will wear an activity monitor on their wrist and keep track of their nightly sleep schedule to establish baseline measures. This will continue for 2 weeks. During the second week of wearing this watch the participant will be asked to come in for a sleep study. This study will consist of two initial nights in the sleep lab and then two more nights in the lab a week later. Participants will be able to leave during the day. Upon completing the sleep assessment, participants will receive bupropion twice daily for 8 weeks. Upon completion of this 8-week treatment, participants will be interviewed to assess the effectiveness of the treatment. One follow-up meeting will occur 6 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder and/or dysthymic disorder

Exclusion Criteria:

* Current treatment with antidepressant drugs
* Major medical illness
* Diagnosis of anorexia nervosa or manic-depressive illness
* Pregnancy

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 130 (Estimated)
Dates: Start 2004-06; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Reduction in depressive symptoms | Measured at Week 8 and Month 6 post-treatment

SECONDARY OUTCOMES:
Improvement in quality of life | Measured at Week 8 and Month 6 post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Uma Rao, MD, Principal Investigator — Meharry Medical Collegey
Locations (1):
- Meharry Medical College, Nashville, Tennessee, United States